CLINICAL TRIAL: NCT01268033
Title: A Prospective, Randomized, Double Blind, Placebo-controlled Phase II/III Study Evaluating the Efficacy of Rituximab in the Prevention of Relapse of Calcineurin Inhibitors Dependent Idiopathic Nephrotic Syndrome of Childhood
Brief Title: Efficacy of Rituximab For the Treatment of Calcineurin Inhibitors Dependent Nephrotic Syndrome During Childhood
Acronym: NEPHRUTIX
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I08013
Record Dates: First submitted 2010-12-15; First posted 2010-12-29 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Childhood Idiopathic Nephrotic Syndrome
Keywords: rituximab; idiopathic nephrotic syndrome; minimal change disease; focal and segmental glomerulosclerosis
MeSH Terms: conditions — Nephrotic Syndrome; Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab (Experimental): two infusions of Rituximab - at the dose of 375 mg/m²
  Interventions: Drug: Rituximab
- placebo (Placebo Comparator): two infusions of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — two infusions - at the dose of 375 mg/m²- will be administered at one week of interval
  Arms: Rituximab
Drug: Placebo — two infusions - at the dose of 375 mg/m² - will be administrered at one week of interval
  Arms: placebo

SUMMARY:
Background

Idiopathic nephrotic syndrome is a rare disease beginning during childhood and treated with immunosuppressants (i.e. steroids, mycophenolate mofetil, cyclophosphamide, cyclosporine).

Renal function of patients suffering from severe, steroid-dependent nephrotic syndrome with failure or toxic side effects of other immunosuppressant treatments is a major matter of concern.

Cyclosporine endangers renal parenchyma (fibrosis) in these patients who must take this treatment for years. At the same time, low doses of cyclosporine allow proteinuria to reappear, which provokes degradation of renal function by focal segmental glomerulosclerosis. Some recent data lead to the conclusion that Rituximab may be effective in such a disease, with a cyclosporin sparing effect.

Purpose

The aim of the study is to evaluate the efficacy of Rituximab versus placebo in the treatment of pediatric patients suffering from severe cyclosporine-dependent nephrotic syndrome.

Abstract Patients will be included in the study in a period of remission of proteinuria. Two infusions of Rituximab - at the dose of 375 mg/m²- or placebo will be administered at one week of interval. Other immunosuppressant treatments will be gradually tapered off with the same tapering pattern in both groups. In case of relapse of nephrotic syndrome, the blinding code will be broken. Rituximab will then be infused to patients having received placebo.

DETAILED DESCRIPTION:
After infusions of Rituximab or placebo, patients will be examined by their nephrologist on a monthly basis during five months. Follow up will be focused on proteinuria, albuminemia, lymphocyte phenotyping and Rituximab pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients over 2 and under 18 years, with an idiopathic nephrotic syndrome (NS)
* Steroid Sensitive Nephrotic Syndrome (according to the French pediatric protocol).

NEPHRUTIX

* Calcineurin inhibitor Dependent NS or NS for which anticalcineurin treatment has not been effective. Others immunosuppressive treatments (MMF) must have failed to control the disease activity.
* Effective contraception for girls of childbearing age.
* The patient is able to understand and has signed a written informed consent OR the parent or legal guardian is able to understand and has signed a written informed consent, which must be obtained prior to the initiation of any study procedure

Exclusion Criteria:

* Terminal renal failure requiring dialysis/transplantation
* Transcutaneous oxygen stauration < 97%
* Clinical or Radiological brochopulmonar or pleural abnormality
* Asymptomatic carrier of Hepatitis B virus our history of Hepatitis B
* Contraindication to Rituximab (RTX)
* Parents/patient refusing to participate in the study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2010-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Proteinuria with relapse of nephrotic syndrome (Serum albumin < 30 g/L) within 5 months | 5 months
  Proteinuria with relapse of nephrotic syndrome (Serum albumin < 30 g/L) within 5 months

SECONDARY OUTCOMES:
- dosing of rituximab for toxicity during and/or after infusion | 5 months
  - toxicity during and/or after infusion
- dosing of rituximab for pharmacokinetics | 5 months
  - dosing of rituximab for pharmacokinetics
- dosing of lymphocyte | 5 months
  - lymphocyte phenotyping
Pediatric Quality of life inventory | 5 months
  Pediatric Quality of life inventory

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GUIGONIS, MD, Principal Investigator — CHU Limoges
Locations (24):
- Queen Fabiola Universitary Children's Hospital, Brussels, Brussels Capital, Belgium
- France (23):
  - Chu Amiens, Amiens, Amiens
  - Chu Besancon, Besançon, Besancon
  - Chu Bordeaux, Bordeaux, Bordeaux
  - Chu Brest, Brest, Brest
  - CHU CAEN, Caen, Caen
  - Chu Clermont Ferrand, Clermont-Ferrand, Clermont Ferrand
  - Chu Grenoble, Grenoble, Grenoble
  - Chu Lille, Lille, Lille
  - Chu Limoges, Limoges, Limoges
  - AP-HM - Hôpital La Timone, Marseille, Marseille
  - Chu Montpellier, Montpellier, Montpellier
  - Chu Nantes, Nantes, Nantes
  - CHU NICE, Nice, Nice
  - AP-HP - Hôpital Necker, Paris, Paris
  - AP-HP - Hôpital Trousseau, Paris, Paris
  - CHU REIMS - American Memorial Hospital, Reims, Reims
  - Chu Rennes, Rennes, Rennes
  - Chu Rouen, Rouen, Rouen
  - Chu Saint Etienne, Saint-Etienne, Saint Etienne
  - Chu Strasbourg, Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse, Toulouse
  - Chu Tours, Tours, Tours
  - Chu Nancy, Vandœuvre-lès-Nancy, Vandoeuvre Les Nancy

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526